CLINICAL TRIAL: NCT01032304
Title: The Efficacy and Safety of Erdosteine in the Long-term Therapy of Chronic Obstructive Pulmonary Disease (COPD). A 12-month, Randomised, Double-blind, Placebo-controlled, Parallel Group, Multicenter Study
Brief Title: The Efficacy and Safety of Erdosteine in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: RESTORE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Edmond Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERD-01-08/EP
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — erdosteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erdosteine (Experimental): 600 mg/day for 12 months
  Interventions: Drug: Erdosteine
- Placebo (Placebo Comparator): Placebo for 12 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erdosteine — One 300 mg capsule twice a day
  Arms: Erdosteine
Drug: Placebo — One capsule twice a day
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of erdosteine, compared to placebo, on exacerbation rate over a 12-month treatment period in patients with moderate-to-severe COPD. Moreover, the effects of erdosteine on pulmonary function parameters, clinical symptoms and quality of life, and the long-term safety of the drug will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* COPD stage II-III GOLD
* At least 2 exacerbations in the previous 2-12 months

Exclusion Criteria:

* Acute exacerbations in the 2 months prior to enrolment
* Diagnosis of asthma and/or other relevant lung diseases
* COPD stage IV
* Unstable concurrent diseases

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Estimated)
Dates: Start 2009-08; Primary Completion 2014-03 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
number of acute exacerbations | 12 months

SECONDARY OUTCOMES:
spirometry parameters | 12 months
COPD symptoms | 12 months
Quality of life | 12 months
Safety and tolerability of erdosteine | 12 months

CONTACTS AND LOCATIONS:
Locations (46):
- Campus Gasthuisberg Dep.t Longfunctiemetingen, Leuven, Belgium
- Bulgaria (4):
  - ASMOH-MC "Sveti Panteleiomon", Sofia
  - Clinic for emergency Medicine and Intensive care, Pneumology and Physiatry, Sofia
  - Clinic of Pulmonary Disease-Military Medical Academy, Sofia
  - Clinical of Pneumology and Physiatry, Varna
- Czechia (9):
  - Plicnì Ordinace, Havlìckuv Brod
  - Poliklinica Moravsky Krumlov, Moravský Krumlov
  - Department of Respiratory Medicine, Faculty Hospital, Olomouc
  - Lipa Centrum Nove Butovice, Prague
  - Lerymed spol. s.r.o., Prague
  - Plicnì Ambulance, Prostějov
  - Plicnì M.I.O., spol. s.r.o., Příbor
  - Plicnì Ordinace, Strakonice
  - Nemonice Znojmo, Znojmo
- Department of Respiratory Diseases, Copenhagen University Hospital, Hvidovre, Denmark
- France (2):
  - Service de Pneumologie, Hopital Bichat, Paris
  - Service de Pneumologie, Hopital Bois-Guillaume, Rouen
- Italy (10):
  - UOC Pneumologia Riabilitativa INRCA, Casatenovo, Lecco
  - UOC di Pneumologia-Ospedale Mater Salutis, Legnago, Verona
  - Dip. Pneumologia Osp. G. Rummo, Benevento
  - U.O. Pneumologia, Bussolengo
  - UOC di Pneumologia- Ospedale Civile di Massa e Carrara, Carrara
  - Ospedale Careggi, Malattie dell'Apparato Respiratorio, Florence
  - UOC Pneumologia Osp. Vito Fazzi, Lecce
  - U.O. Pneumologia, Macerata
  - UO di Pneumologia Osp. San Paolo, Milan
  - Ospedale San Carlo Borromeo, Dipartimento Broncocardiopneumologico, Milan
- Poland (6):
  - Szpital Uniwersytecki 2, Bydgoszczy
  - Klinika Pulmonologii II Katedry, Collegium Medicum Uniwersytetu, Krakow
  - Katedra Pulmunologii i Alergologii, Klinika Gruźlicy Uniwersytetu Medycznego, Lodz
  - Katedra i klinika Pulmonologii, Uniwersytet Medyczny, Poznan
  - NZOZ "Darmeticus", Warsaw
  - Katedra i Klinika Pneumonologii, Warszawski Uniwersytet Medyczny, Warsaw
- Romania (6):
  - Institutul de Pneumoftiziologie "Marius Nasta", Bucharest
  - Novo Medica, Bucharest
  - Spitalul de Pneumoftiziologie "Leon Daniello", Cluj-Napoca
  - Spitalul Clinic de Pneumoftiziologie, Iași
  - Clinica Pneumologie I, Spitalul Clinic Judetean Mureş, Târgu Mureş
  - Spitalul de Pneumoftiziologie "Victor Babes", Timișoara
- Slovakia (4):
  - Nemocnica s Poliklinicou "Svateho Jakuba"n.o., Bardejov
  - Inspiro, Humenné
  - Specializovana NemocnicaSvorada Zobor n.o., Nitra
  - Narodny Ustav Tuberculozy, Vyšné Hágy
- United Kingdom (3):
  - Regional Respiratory Centre, Belfast City Hospital, Belfast
  - Cardiovascular and Respiratory Studies Department, Hull
  - Aintree Chest Centre, University Hospital Aintree, Liverpool

REFERENCES:
- [Derived] Dal Negro RW, Wedzicha JA, Iversen M, Fontana G, Page C, Cicero AF, Pozzi E, Calverley PMA; RESTORE group; RESTORE study. Effect of erdosteine on the rate and duration of COPD exacerbations: the RESTORE study. Eur Respir J. 2017 Oct 12;50(4):1700711. doi: 10.1183/13993003.00711-2017. Print 2017 Oct. PMID 29025888